CLINICAL TRIAL: NCT05985356
Title: Neuromodulation for Comorbid Hoarding Disorder and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Elizabeth Twamley, Professor of Psychiatry, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG106837
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Hoarding Disorder; Hoarding; Depression
Keywords: TMS; Transcranial magnetic stimulation
MeSH Terms: conditions — Hoarding Disorder; Hoarding; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- iTBS (Experimental): intermittent Theta Burst Stimulation (a form of transcranial magnetic stimulation) targeting the left dorsolateral prefrontal cortex
  Interventions: Device: iTBS

INTERVENTIONS:
Device: iTBS — iTBS targeting the left dorsolateral prefrontal cortex; 20 sessions over 4 weeks.
  Other Names: rTMS

SUMMARY:
The primary goal of this study is to evaluate whether intermittent theta burst stimulation (iTBS) is effective for treating depression in people who have depression and chronic hoarding disorder (HD). The study will also evaluate whether this treatment can improve HD symptoms, cognitive performance, and brain region connectivity. The study team will investigate how the treatment works for depression, as well as other factors that can enhance or hinder treatment, such as pre-treatment level of depression, cognitive performance, or brain region connectivity.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male, female, or non-gender conforming individuals (i.e. those who do not identify as male or female)
4. All racial and ethnic groups
5. Ages 18 to 70
6. Meets criteria for current Major Depressive Episode within the context of Major Depressive Disorder, per HAM-D and DIAMOND.
7. Meets criteria for current Hoarding Disorder, per SIHD
8. Score of 18 or higher on the HAMD-17, indicating moderate to severe depressive symptoms
9. Stable on psychiatric medications for 6 weeks, with no changes to psychiatric medications expected during the study period
10. No contraindications to TMS (passes the TMS Adult Safety Screening questionnaire)
11. No contraindications to MRI (passes MRI safety screening questionnaire)
12. Able to commit to the treatment schedule
13. Able to complete assessment procedures in English
14. Intact decision-making capacity and ability to provide voluntary informed consent

Exclusion Criteria:

1. History of other neurological condition including but not limited to: conditions associated with increased intracranial pressure; space occupying brain lesions; cerebral aneurysm; stroke; transient ischemic attack within past two years; Parkinson's disease; Huntington's disease; dementia; multiple sclerosis; history of brain surgery; epilepsy; seizure except those therapeutically induced by electroconvulsive therapy (ECT) or a febrile seizure of infancy
2. Implanted medical devices that are not explicitly recognized as MRI safe, including cardiac pacemaker, medication pump, aneurysm clip, shunt, stimulator, cochlear implant, electrodes, or any other metal object within or near the head (excluding the mouth) that cannot be safely removed
3. Active manic or psychotic illness per DIAMOND
4. Current substance use disorder per DIAMOND
5. Current active suicidal or spontaneously disclosed homicidal ideation. Active suicidal ideation for this study is defined as a score of 3 or greater on the HAMD-17 and/or 3 or more on the PHQ-9.
6. Pregnant or intending to become pregnant within the study period; breastfeeding
7. Other sensory conditions or illnesses precluding participation in assessments or treatment
8. Current dose of lorazepam 2 mg or greater daily (or benzodiazepine equivalent) or any anticonvulsant due to the potential to limit iTBS efficacy
9. Taking medication that lowers seizure threshold
10. Previous failed treatment with rTMS, iTBS, or ECT

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Savings Inventory -- Revised | change from baseline to 8 weeks
  self-reported symptoms of hoarding disorder
Hamilton Rating Scale for Depression | change from baseline to 8 weeks
  depression symptom severity

SECONDARY OUTCOMES:
Hoarding Rating Scale | change from baseline to 8 weeks
  self-reported symptoms of hoarding disorder
Patient Health Questionnaire - 9 | change from baseline to 8 weeks
  self-reported symptoms of depression
Neuropsychological Global Deficit Score | change from baseline to 8 weeks
  neurocognition composite
resting state functional connectivity | change from baseline to 4 weeks
  connectivity between subgenual nucleus accumbens and dorsolateral prefrontal cortex as measured by functional magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Twamley, PhD, Principal Investigator — UC San Diego
Locations (1):
- UC San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
Data can be de-identified and made available upon request.